CLINICAL TRIAL: NCT02614274
Title: Pilot Assessment of the Biochemical Response of a Novel Nutraceutical Joint Health Formulation Using a Multiplexed Biomarker Approach
Brief Title: Nutramax Joint Health Formulation Biochemical Response Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Nutramax Laboratories, Inc. (Industry)
Responsible Party: Principal Investigator, James Cook, DVM, PhD, OTC, Director, Comparative Orthopaedic Laboratory, Orthopaedic Research Division & Mizzou BioJoint Center, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1213242
Record Dates: First submitted 2015-11-24; First posted 2015-11-25 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-04

CONDITIONS: Osteoarthritis, Knee
Keywords: knee; pain; osteoarthritis; nutraceutical; nutrition; supplement; non-surgical; biomarker; joint health
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutraceutical joint health formulation (Experimental): A Proprietary Blend
  Interventions: Dietary Supplement: Nutraceutical joint health formulation

INTERVENTIONS:
Dietary Supplement: Nutraceutical joint health formulation — A Proprietary Blend

SUMMARY:
The Nutramax test article is a nutritional supplement that contains several ingredients shown to potentially provide benefit to patients suffering from a painful and sometimes debilitating condition of the knee called "osteoarthritis."

This is a pilot study that is intended to determine whether results from a proprietary testing panel conducted on blood and urine samples will correlate with data from physical examination and validated surveys that measure participants' quality of life and physical capabilities.

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the knee is a significant source of morbidity, especially in patients over the age of 40 and is associated with more than $90 billion in US health care costs annually. While a myriad of clinical interventions are available, the mainstays of OA therapy are the NSAIDs, a class of compounds with well documented side effects including death; the risks of which increase with patient age and chronic use. Assessing the effectiveness of OA treatment modalities is often complicated by a high placebo effect, making purely clinical assessment of outcomes difficult. It is therefore desirable to develop an objective assessment tool for both the diagnosis/staging of knee OA and patient response to interventional therapies.

Participants in this study will receive a formulation of the nutraceutical (test article). They will be asked to take 3 pills at once per day for 40-44 days. There will be either 4 or 5 study visits. If participants have been using certain medications or dietary supplements, they will be asked to return one week from the initial screening, making a total of 5 visits in the study. If they have not been using key medications or dietary supplements, then study activities will begin on the day of the initial screening and they will only have 4 study visits.

Participants will be asked to complete a series of questionnaires about their health, and have their blood drawn (15 mls or about 3 teaspoons), and provide a urine sample at 4 visits. In addition, at the first visit, we will collect information from participants' medical record and they will have a physical exam.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to understand and sign the informed consent.
2. Subject is willing and able to comply with the protocol.
3. Male or female subjects of any race, aged 40 to 64 years
4. Subject has a BMI of 24 to 40 kg/m2
5. Subject has had pain in one or both knees for a minimum of 15 days within the 30 days prior to the start of the study.
6. Subject has had symptoms of knee pain for at least 6 months.
7. Subject has been diagnosed within the previous 30 days with moderate to severe knee osteoarthritis - based on attending physician's diagnosis from physical exam in conjunction with Kellgren-Lawrence X-ray grade of ≥ 2 (radiographs taken within previous 30 days must be available to the investigator, or be obtained at the screening visit).
8. Subject can walk.
9. Before study enrollment, subject routinely uses acetaminophen (at any dose) with a history of therapeutic benefit.
10. Subject has a visual analogue scale (VAS) score of ≥ 4 at the initial visit. Subject may continue taking acetaminophen at the screening but will not have taken additional analgesics for at least 48 hours prior to the initial visit.
11. Female subject abstains from sexual intercourse, is surgically sterile, post-menopausal, or agrees to use a FDA-approved method of birth control.

Exclusion Criteria:

1. Subject has any of the following medical conditions:

   1. active heart disease - defined as currently under the care of a cardiologist
   2. high blood pressure (≥ 140/90 mmHg)
   3. renal or hepatic impairment/disease
   4. Type I or II diabetes
   5. Bipolar or major depressive disorder or a history of other psychiatric illness requiring hospitalization in the past 6 months.
   6. Parkinson's disease
   7. unstable thyroid disease
   8. immune disorder (such as HIV/AIDS)
   9. multiple sclerosis or any other autoimmune disorder
   10. any arthritic condition, other than OA, affecting a joint other than the knee
   11. acute septic arthritis
   12. fibromyalgia or other chronic pain syndromes (OA in locations other than knee allowed)
   13. gout and hyperuricemia
   14. peptic ulcer disease and/or history of upper gastrointestinal bleeding
   15. any medical condition deemed exclusionary by the Principal Investigator (PI)
2. Subject has a history of cancer (except localized skin cancer without metastases or in situ cervical cancer) within five years prior to screening.
3. Subject has had a significant injury to the target joint within the past 12 months.
4. Subject plans to have knee surgery in the next 2 months.
5. Subject has had an asthma attack, hives, or other allergic reaction with aspirin or any other NSAID medication.
6. Subject has an allergy to avocados, soybeans, shellfish or any other ingredient in the test product.
7. Subject requires additional analgesic or a change from acetaminophen. (Subjects requiring acetaminophen dose adjustments may remain in the study and all such dose and/or schedule changes shall be recorded in the raw data and daily patient diary).
8. Subject is currently taking any medication or suffers from a medical condition, deemed to potentially interfere with the objectives of the study as determined by the PI.
9. Subject has a history of drug or alcohol abuse in the past 12 months.
10. Subject is currently consuming more than 2 standard alcoholic beverages a day. A standard alcoholic beverage is defined as 12 ounces of beer, 5 ounces of wine, or 1.5 ounces of liquor.
11. Subject does not agree to use a FDA-approved method of birth control or is pregnant, lactating, or planning to become pregnant during the study period.
12. Subject has any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the subject or the quality of the study data.
13. Subject is participating or has participated in another research study within 30 days prior to screening.
14. Subject has used, or intends to use, any oral or injectable NSAID (e.g., ketorolac, aspirin, ibuprofen, naproxen, diclofenac, etc.) within 7 days prior to screening through study completion.
15. Subject has been treated with oral corticosteroids within 4 weeks prior to screening.
16. Subject had intra-articular corticosteroids in the target joint within 3 months prior to screening.
17. Subjects may not take any dietary, vitamin, mineral, or herbal supplements within 7 days prior to Day 0 through study completion. For subjects taking such products at time of the initial visit, a seven-day washout period prior to study Day 1 is allowed EXCEPT for joint health/anti-inflammatory products (see # 18).
18. Subjects who are currently taking or have taken for ≥ 30 consecutive days OR ≥ 60 days total, within the 180 days prior to screening, dietary products intended to decrease inflammation, body pain and/or improve joint health; including, but not necessarily limited to, glucosamine, chondroitin, avocado-soybean unsaponifiable (ASU), and methylsulfonylmethane (MSM) shall be excluded from the study.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Cook, DVM PhD OTC, Principal Investigator — University of Missouri, Missouri Orthopaedic Institute
Locations (1):
- University of Missouri, Missouri Orthopaedic Institute, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nutraceutical Joint Health Formulation: A Proprietary combination of Glucosamine HCl, Chondroitin Sulfate, Avocado/Soybean Unsaponifiables (ASU), and 3-O-Acetyl-11-Keto β-Boswellic Acid (AKBA)
Period: Overall Study
Arm/Group | Nutraceutical Joint Health Formulation
Started | 9
Completed | 5
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Nutraceutical Joint Health Formulation
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Serum Biomarkers
Description: Blood will be assessed using a proprietary panel of biomarkers of inflammation. Blood and urine were collected, processed, and analyzed using a proprietary panel of biomarkers using the Luminex system as previously described (Garner, et al; Roller, et al). In addition, serum hsCRP was analyzed.
Time Frame: 42 days
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Nutraceutical Joint Health Formulation
Number analyzed (Participants) | 5
pg/ml
  PGE2 | 130 (17)
  MMP1 | 114 (48)
  GRO | 109 (63)
  IL8 | 63 (3)
  hsCRP | 14 (1)

2. Primary Outcome: Urine Biomarkers
Description: Urine will be assessed using a proprietary panel of biomarkers of inflammation.
Time Frame: 42 days
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Nutraceutical Joint Health Formulation
Number analyzed (Participants) | 5
pg/ml
  PGE2 | 7.9 (5.8)
  MMP2 | 17.2 (10)
  MMP3 | 3.2 (3)
  GRO | 2.9 (2.9)
  IL8 | 1 (1)

3. Secondary Outcome: Patient Reported Quality of Life Via SF-36 (36-Item Short Form Health Survey) Improvement
Description: The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software.
  Mean+-SD among of improvement is reported.
Time Frame: 42 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nutraceutical Joint Health Formulation
Number analyzed (Participants) | 5
units on a scale
  Physical Function | 70 (30.8)
  Role limitations due to physical health | 50 (54.8)
  Role limitations due to emotional problems | 80 (44.7)
  Energy/fatigue | 70 (11)
  Emotional well being | 77.6 (11.1)
  Social functioning | 92.5 (12.4)
  Pain | 71 (15.9)
  General health | 81 (24.9)

4. Secondary Outcome: Patient Reported Opinions (About Their Knee) Via KOOS (Knee Injury and Osteoarthritis Outcome Score)
Description: Knee injury and Osteoarthritis Outcome Score (KOOS). A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Time Frame: 42 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nutraceutical Joint Health Formulation
Number analyzed (Participants) | 5
units on a scale
  Symptoms | 44.3 (23.1)
  Pain | 50.6 (19.4)
  Activities of Daily Living | 60 (15.1)
  Sports | 37 (23.9)
  Quality of Life | 30 (28.4)

5. Secondary Outcome: Patient Reported Survey to Assess: Pain, Stiffness, and Physical Function in Patients With Hip and/or Knee Osteoarthritis (OA) Via WOMAC (Western Ontario and McMaster Universities Arthritis Index)
Description: The Western Ontario and McMaster Universities Arthritis Index (WOMAC). A lower score indicates less severe symptoms, a higher score indicates more severe symptoms. The range of scores as is follows: 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Function.
Time Frame: 42 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nutraceutical Joint Health Formulation
Number analyzed (Participants) | 5
units on a scale
  Pain | 10.8 (5.6)
  Stiffness | 3.6 (2.2)
  Function | 26.4 (13.6)

6. Secondary Outcome: Patient Reported Survey to Assess Symptoms and Function in Daily Living Via IKDC (International Knee Documentation Committee) Subject Exam
Description: International Knee Documentation Committee (IKDC). Each subscale is scored from 0-100, with 100 being no limitation with activities of daily living or sports activities and the absence of symptoms.
Time Frame: 42 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nutraceutical Joint Health Formulation
Number analyzed (Participants) | 5
units on a scale
  Symptoms | 56.8 (29.1)
  Sports | 57 (26.4)
  Function | 52 (34.4)

ADVERSE EVENTS:
Arm/Group | Nutraceutical Joint Health Formulation
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nutraceutical Joint Health Formulation (N=9)
headache (Nervous system disorders) | 1 (1) — episode of headache and a generalized viral infection such as influenza, treated and ibuprofen and resolved completely. Unrelated but still removed from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No